CLINICAL TRIAL: NCT05308511
Title: A Prospective, Multi-center, Randomized and Self-controlled Clinical Trial to Evaluate the Effectiveness and Safety of Colon Capsule Endoscope System for Capturing and Viewing Colon Images Clinically
Brief Title: Evaluating the Effectiveness and Safety of Colon Capsule Endoscope System for Capturing and Viewing Colon Images
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Collaborators: Renmin Hospital of Wuhan University (Other); Beijing Tsinghua Changgeng Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: AK-CTP-01
Record Dates: First submitted 2022-03-14; First posted 2022-04-04 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2022-04

CONDITIONS: Prospective Study

STUDY DESIGN:
Intervention Model Description: The trial is a prospective, multi-center,randomized, self-controlled,and non-inferiority design clinical trial. Subjects included in the research were subject to capsule endoscopy in one swallowing order (two in total), which was determined by the pre-generated random number.
  Swallowing order I: First swallow the trial device(PC-I) for examination, and then swallow the comparator device(COLON2) for examination at an interval of 2h.
  Swallowing order II: First swallow the comparator device(COLON2) for examination, and then swallow the trial device(PC-I) for examination at an interval of 2h.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Swallowing order I (Experimental): First swallow the trial device(PC-I) for examination, and then swallow the comparator device(COLON2) for examination at an interval of 2h.
  Interventions: Device: PC-I and COLON2
- Swallowing order II (Experimental): First swallow the comparator device(COLON2) for examination, and then swallow the trial device(PC-I) for examination at an interval of 2h.
  Interventions: Device: COLON2 and PC-I

INTERVENTIONS:
Device: PC-I and COLON2 — First swallow the trial device(PC-I) for examination, and then swallow the comparator device(COLON2) for examination at an interval of 2h.
  Arms: Swallowing order I
Device: COLON2 and PC-I — First swallow the comparator device(COLON2) for examination, and then swallow the trial device(PC-I) for examination at an interval of 2h.
  Arms: Swallowing order II

SUMMARY:
The trial is a prospective,multi-center, randomized and self-controlled clinical trial. The research plan will be implemented in a clinical trial center with the qualification of clinical trial agency, and 128 subjects will be planned to be included. Subjects signing the Informed Consent Form, meeting the trial conditions and all inclusion criteria and failing to meet any exclusion criteria will be included in the research. The trial device was Colon Capsule Endoscope System for colonoscopy(PC-I) manufactured by ANKON Technologies Co.,Ltd. while the comparator device was Capsule Endoscopy System(PillCam COLON2) manufactured by Given Imaging Inc. The main evaluation indicator is the excellent rate of image quality, while secondary evaluation indicators are the consistency rate of lesion detection, completion rate of colonoscopy, discharge time of capsule endoscopy, colon passing time and device performance evaluation. Safety evaluation indicators include adverse events(or Serious adverse events), device-related adverse events(or Serious adverse events) and device defects. In the end, the effectiveness and safety of Colon Capsule Endoscopy diagnostic system manufactured by ANKON Technologies Co.,Ltd. for capturing and viewing colon images clinically were verified according to the above indicator results.

DETAILED DESCRIPTION:
According to the relevant requirements of Standard for Quality Management of Medical Device Clinical Trials (Order No. 25 of the National Health and Family Planning Commission of the People's Republic of China of China Food and Drug Administration), the sample size was estimated based on the excellent rate of the image quality of the main endpoint by referring to the domestic and foreign literatures using positive comparator devices. Combined with literatures and comments of clinical experts, the research set the excellent rate of image quality of comparator device Ps as 95%, and estimated the excellent rate of image quality of trial device Pt as 95%. In the research, the non-inferiority trial design was adopted, with α = 0.025 (unilateral), assurance 1 - β = 0.8, and non-inferiority boundary value of -10%, and self-control was adopted. It is assumed that the redundant parameter (that is, the proportion of subjects whose evaluation results of image quality between trial devices and comparator devices are inconsistent) was 0.095 (that is, Pt (1 - Ps) + Ps (1 - Pt)), the total sample size of the two groups was 102 cases calculated by PASS2021, with 51 cases in each swallowing orders I and II. Considering the shedding and rejection rate of 20% during the trial, a total of 128 subjects were needed, with 64 cases in each swallowing orders I and II.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old (including 18 years old), male or female;
* Subjects intending to take capsule endoscopy and/or the electronic endoscopy of the lower digestive tract;
* The subject signed the ICF voluntarily.

Exclusion Criteria:

* Subjects suffering from swallowing obstruction or deglutition disorders;
* Subjects who underwent gastrointestinal abdominal surgery in the past 6 month (except for simple surgery unlikely to cause intestinal obstruction according to the clinical judgment of researchers).
* Subjects of CRC (advanced adenomatous polyp and CRC) failing to undergo the surgery;
* Subjects suffering from gastrointestinal obstruction, stenosis or fistula;
* Subjects being unable to take capsule endoscopy due to intestinal preparation failure;
* Subjects with cardiac pacemakers or other implantable electronic medical devices;
* Subjects failing to meet requirements for the abdominal surgery or refusing to take any abdominal surgery;
* Female subjects during pregnancy, lactation or having a pregnancy plan recent 3 months;
* Subjects who underwent colonoscopy within 2 years, with the negative result;
* Subjects suffering from type 1 or type 2 diabetes;
* Subject taking incomplete colonoscopy due to enteropathy of severe ulcerative colitis, radiation enteritis or non-steroidal anti-inflammatory drugs[4];
* Subjects suffering from any disease considered to increase the retention risk of the capsule endoscopy;
* Subjects currently participating in another clinical trial of drugs or devices;
* Other circumstances unsuitable for inclusion upon judgment by the researcher.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-08-04 (Actual)

PRIMARY OUTCOMES:
The excellent rate of image quality. | 1 day
  The main effectiveness evaluation indicator is the excellent rate of image quality, which is for the statistics of the difference between the excellent rate of image quality of trial devices and comparator devices and unilateral 97.5% confidence interval. If the lower limit of unilateral 97.5% confidence interval of the difference between the two groups is greater than -10% of the non-inferiority boundary value, it can be considered that the excellent rate of image quality of trial devices is not inferior to that of comparator devices.

SECONDARY OUTCOMES:
The consistency rate of lesion detection | 1 day
  2 associate chief physicians of digestive endoscopy or attending physicians with more than 5 years of endoscopic experience adopted independent film reading in the center for recording of the lesion detection in the image through back-to-back interpretation and analysis. Then record the number of lesions detected consistently.
Completion rate of colonoscopy | 1-14 days
  Colonoscopy is completed before the battery runs out, and the capsule endoscopy captures the rectal segment image or the image that the capsule endoscopy is discharged from the body.
Discharge time of capsule endoscopy | 1-14 days
  The discharge time of the capsule endoscopy is from swallowing capsule endoscopy to discharging capsule endoscopy.
Colon passing time | 0.5-10hours
  Colon passing time is from the capsule endoscopy's arrival at the ileocecal valve to the capsule endoscopy's discharge from the body.
Device performance evaluation | 1day
  Subjective evaluation of the performance of the trial and control devices.

CONTACTS AND LOCATIONS:
Overall Officials: XiaoHua Hou, MD.PhD, Principal Investigator — Union Hospital of Tongji Medical College of Huazhong University of Science and Technology
Locations (1):
- Union Hospital of Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei, China